CLINICAL TRIAL: NCT06300801
Title: Postoperative Pancreatic Fistula in Patients Undergoing Pancreaticoduodenectomy
Acronym: popf
Status: No longer available | Type: Expanded Access
Sponsor: Erol Olcok Corum Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Bahadır Kartal, Principal Investigator, Erol Olcok Corum Training and Research Hospital
Other Study IDs: 2023-48; hitit (Other: hitit university)
Record Dates: First submitted 2024-02-16; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-02

CONDITIONS: Pancreatic Fistula After Pancreaticoduodenectomy; C-Reactive Protein; Albumin
Keywords: albumin; pancreatic fistula; c- reactive protein
MeSH Terms: conditions — Pancreatic Fistula

INTERVENTIONS:
Diagnostic Test: Is the preoperative c-reactive protein/albumin ratio successful in predicting postoperative pancreatic fistula in patients undergoing pancreatoduodenectomy? — In this study, predicting pancreatic fistula before surgery will reduce postoperative complications and mortality.

SUMMARY:
Pancreaticoduodenectomy (PD) is a complex procedure performed in patients with malignant or benign tumors of the pancreatic head and periampullary region, associated with high morbidity and mortality. Postoperative pancreatic fistula (POPF) is the most common and clinically significant complication following PD. In this study, the investigators aim to predict pancreatic fistula using the C-reactive protein-albumin ratio (CAR). The total number of participants expected to be included in this research comprises patients who underwent PD between 2017 and 2023 and developed pancreatic fistula. The participants invitation is based on the detection of a pancreatic fistula. This study is conducted for research purposes and participation is voluntary. No interventions will be performed on the participants as part of this study; however, we have prepared this form to obtain participant permission to gather certain information. If the participants consent to the use of information for scientific purposes with the guarantee of confidentiality, they will be asked to sign a consent form.

DETAILED DESCRIPTION:
Pancreaticoduodenectomy (PD) is a complex procedure performed in patients with malignant or benign tumors of the pancreatic head and periampullary region, associated with high morbidity and mortality rates. Despite dramatic advancements in surgical techniques and perioperative management, reported morbidity and mortality rates following PD are 41.56% and 2.88%, respectively, which remain unsatisfactory. Postoperative pancreatic fistula (POPF) is the most common and clinically significant complication following PD. Therefore, accurate and timely prediction of POPF after PD is necessary to reduce secondary mortality from serious complications and optimize individual patient treatment decisions. The C-reactive protein-albumin ratio (CAR) is an inflammatory marker calculated by dividing serum CRP levels by albumin levels and has been associated with poor prognosis in sepsis patients. This study aimed to investigate the predictive significance of CAR for POPF.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 80 years
* Diagnosed with pancreatic cancer
* Patients without recurrence

Exclusion Criteria:

* Patients who underwent total pancreatectomy
* Data were not available
* Patients outside the specified age range

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Hitit University Erol olçok Traning and research Hospital, Çorum, Merkez
  - Hitit University Erol olçok Traning and resourge Hospital, Çorum, Merkez

REFERENCES:
- [Background] Sakamoto T, Yagyu Y, Uchinaka EI, Morimoto M, Hanaki T, Tokuyasu N, Honjo S, Fujiwara Y. Predictive Significance of C-reactive Protein-to-albumin Ratio for Postoperative Pancreatic Fistula After Pancreaticoduodenectomy. Anticancer Res. 2019 Nov;39(11):6283-6290. doi: 10.21873/anticanres.13838. PMID 31704858